CLINICAL TRIAL: NCT03847675
Title: "Reach Out and Read" Arabic to Promote Parental Reading to Toddlers and Preschoolers
Brief Title: Reach Out and Read Arabic to Promote Arabic Literacy in Toddlers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment and lack of funding
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Lama Charafeddine, Associate Professor of Pediatrics and Neonatology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PED.LC.13
Record Dates: First submitted 2019-01-24; First posted 2019-02-20 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-02

CONDITIONS: Child Development
Keywords: Reach out and Read; Arabic literacy; Child development

STUDY DESIGN:
Intervention Model Description: An experimental double blinded parallel arms randomized controlled trial with pre and post-intervention assessment over a period of 12 months with a follow up plan at 2 and 3 years of age
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The research assistant introduces the adapted 'Reach out and Read" program and informs participants about the benefits of reading to children at an early age. A 4:50 minutes video clip would be shown during the initial visit. This video discusses the benefits of reading displaying practical tips for parents; it includes tips on how to read, pointing at the words.
  A schematic pamphlet highlighting the importance of reading Arabic to children and the impact of such reading on children's brain development, vocabulary acquisition and behavior in addition to the impact on the parent child bond and relationship is given to the parents.
  After each visit participants will receive an age appropriate book for their child.
  Focus groups will be conducted by a qualitative researcher
  Interventions: Behavioral: Reach out and Read
- Control (No Intervention): The research assistant gives routine advice on child development including importance of reading and advice on nutrition and safety and gives parents a leaflet about early child development and complementary feeding

INTERVENTIONS:
Behavioral: Reach out and Read — The intervention group will be viewing a video encouraging to read to their children and giving tips on reading methods, in addition will be given a schematic pamphlet highlighting the importance of reading Arabic to children.
  After each visit participants will receive an age appropriate book for their child (a total of 3 books). The first book consist of popular nursery rhymes that are usually sung for younger infants. The choice of the 2 other books is based on recommendations from an early child educator according to age specificity.
  Focus group conducted by a qualitative researcher will follow the protocol reported by Richard A. Krueger.
  Arms: Intervention

SUMMARY:
The goal of this study is to encourage parents to read Arabic books to their children from an early age and by extension children will be more likely to read Arabic books and ultimately improve their Arabic literacy.

The investigators' hypothesis is that an adapted "Reach Out and Read" program will result in an increase in the proportion of parents reading Arabic books to their children after the intervention.

DETAILED DESCRIPTION:
Early reading for toddlers has been linked to a better grasp of the fundamentals of language as they approach school age, as reading exposes the child to rich language and diverse content. Reach Out and Read program (ROR) is an American non-profit organization that advocates for childhood literacy.

In this study the investigators aim to implement an adapted version of the "Reach Out and Read" program and to encourage parents to read Arabic books to their children in order for this to become a daily habit. The goal of this study is to see an increase in the proportion of parents who read Arabic books to their children and by extension children will grow up loving to read Arabic books and ultimately may have improved Arabic literacy.

ELIGIBILITY:
Inclusion Criteria:

* Parents must identify the study's settings as the usual site for their child regular checkups
* Families are eligible if at least one parent understands, speaks and reads Arabic.
* The child's age between 4 and 6 months at the time of the enrollment

Exclusion Criteria:

* Children diagnosed or displaying severe behavioral, cognitive, or physical impairment, that prevents them in meaningfully engaging in a reading activity example: severe autism, profound developmental or intellectual delay.

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of parents reading Arabic books to their children | 3 years
  Measure the proportion of parents reading Arabic books to their children after 3 intervention visits, when their child is about 15 months of age. Parental reading is defined as reading for a minimum of 10 minutes daily for at least 5 days per week.

SECONDARY OUTCOMES:
Weekly frequency of parental reading in Arabic before, and after the intervention | 3 years
  The weekly frequency of parental reading in Arabic before, and after the intervention at each age group (9, 12 and 15 months), then at 2 and 3 years of age as compared between experimental and control group
Children's vocabulary and language / words' | 3 years
  The children's vocabulary and language / words' acquisition in the experimental compared to the control group at 2 years and 3 years.
Children's early developmental milestones | 3 years
  The children's early developmental milestones in the experimental compared to the control group at 2 years and 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Lama Charafeddine, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

REFERENCES:
- [Background] Duursma E, Augustyn M, Zuckerman B. Reading aloud to children: the evidence. Arch Dis Child. 2008 Jul;93(7):554-7. doi: 10.1136/adc.2006.106336. Epub 2008 May 13. No abstract available. PMID 18477693
- [Background] Kuhl PK. Early Language Learning and Literacy: Neuroscience Implications for Education. Mind Brain Educ. 2011 Sep;5(3):128-142. doi: 10.1111/j.1751-228X.2011.01121.x. PMID 21892359